CLINICAL TRIAL: NCT06455228
Title: Long Peripheral Intravenous Catheter Insertion Site and Catheter-related Complications in Antimicrobial Therapy: a Randomized Controlled Trial
Brief Title: Long Peripheral Intravenous Catheter Insertion Site and Catheter-related Complications in Antimicrobial Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-2233-01
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Antimicrobial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper arm (Experimental): ①Evaluation: The puncture site was determined by senior nurses based on group assignment before placement. The depth and diameter of the pre-punctured vein were measured using ultrasound assessment, and the intima of the pre-punctured vein was examined without applying a tourniquet. ②Catheterization: A 3 Fr, 8 cm tip-opened long PIVC was used. Catheters were placed according to the designated sites for each group using ultrasound-guided and accelerated Seidinger techniques. After confirming catheter placement, needleless connectors and extension were attached, and the catheter was secured without tension using a sterile transparent dressing. ③Maintenance: Specialized nurses were trained to monitor and evaluate catheter function daily. Clinical nurses conducted routine maintenance until the study completion. Daily data were recorded and updated in computerized records.
  Interventions: Device: insert catheter
- forearm (Other): ①Evaluation: The puncture site was determined by senior nurses based on group assignment before placement. The depth and diameter of the pre-punctured vein were measured using ultrasound assessment, and the intima of the pre-punctured vein was examined without applying a tourniquet. ②Catheterization: A 3 Fr, 8 cm tip-opened long PIVC was used. Catheters were placed according to the designated sites for each group using ultrasound-guided and accelerated Seidinger techniques. After confirming catheter placement, needleless connectors and extension were attached, and the catheter was secured without tension using a sterile transparent dressing. ③Maintenance: Specialized nurses were trained to monitor and evaluate catheter function daily. Clinical nurses conducted routine maintenance until the study completion. Daily data were recorded and updated in computerized records.
  Interventions: Device: insert catheter

INTERVENTIONS:
Device: insert catheter — A fixed routine for pre-insertion cleaning and equipment was followed, including hand washing, placing the patient in a recumbent position, skin antisepsis, and preparation of the sterile field. Catheter insertion was performed by senior specialized nurses in the intravenous treatment room, which was a standardized setting for venipuncture.

SUMMARY:
This study applies long PIVCs to patients undergoing antimicrobial therapy, and compares the effects of different placement sites, aiming to provide a reference basis for patients undergoing antimicrobial treatment to select the optimal placement site, thus reducing complications, prolonging catheter retention time, and alleviating the patient's pain.

DETAILED DESCRIPTION:
This study investigates the use of long PIVCs in patients undergoing antimicrobial therapy, and compares the effects of different insertion sites. The aim is to provide evidence-based recommendations for the optimal placement site for long PIVCs in antimicrobial treatment, with the goals of reducing complications, prolonging catheter retention time, and alleviating patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* ① estimated time of intravenous infusion ≥1 week; ② age: ≥18 years; ③ antimicrobial therapy was only used for treatment during hospitalization, with a pH value of 5-9 and osmotic pressure < 900 mOsm/L; and ④ patients were conscious and able to communicate normally; ⑤ the catheter-to-vessel ratio is less than 45%.

Exclusion Criteria:

* ① a history of radiotherapy, thrombosis, and trauma at the catheterization site and ② plans to discharge with a catheter during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter-related complications | After insertion of catheter
  Catheter-related complications were assessed including thrombophlebitis, other phlebitis, catheter occlusion, bleeding, catheter-related infections, and weeping.

SECONDARY OUTCOMES:
Puncture success rate with one-attempt | After insertion of catheter
  The puncture success rate with one-attempt refers to the instance where the puncture needle successfully enters the target vein on the first attempt without needing to change the puncture site.
The procedure time | After insertion of catheter.
  The procedure time is defined as the duration from the start of skin disinfection to the stabilization of the catheter with dressing.
Indwelling catheter duration | After insertion of catheter
  The Indwelling catheter duration refers to the number of days between the date of catheter placement and its removal.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Linfang, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao L, Jin X, Li X, Liu C, Wang J, Cao X, Zeng X, Zhuang Y. Differences in catheter-related complications to insertion site selection for long peripheral intravenous catheters in antimicrobial therapy: a randomized controlled trial. BMC Nurs. 2025 Feb 4;24(1):131. doi: 10.1186/s12912-025-02749-y. PMID 39905387